CLINICAL TRIAL: NCT03749291
Title: Effect of a Motivational Intervention on the Gut Microbiota and the Components of the Metabolic Syndrome in a Population of Obese Children
Brief Title: Motivational Intervention on the Gut Microbiota of Obese Children
Acronym: MICROBEkids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Veronica Luque, Dr. PhD, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI18/00226
Record Dates: First submitted 2018-10-08; First posted 2018-11-21 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-05

CONDITIONS: Microbial Colonization
Keywords: Childhood Obesity; Motivational therapy; Dietary Patterns; Cardiovascular disease risk
MeSH Terms: conditions — Communicable Diseases; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obemat2.0 Intervention Group (Experimental): Obese children (BMI >97th percentile of the Spanish curves from Hernández 1988) Ages: 8 to 13 at baseline (9 to 15y at the end of the intervention)
  Interventions: Other: Obemat2.0 therapy
- Control Group (Active Comparator): Obese children (BMI >97th percentile of the Spanish curves from Hernández 1988) Ages: 8 to 13 at baseline (9 to 15y at the end of the intervention)
  Interventions: Other: Usual Clinical Practice

INTERVENTIONS:
Other: Obemat2.0 therapy — Lifestyle (diet & physical activity) structured recommendations through a motivational interview.
  Duration: 12(+3) months Description: 1 visit/month & 3 Workshops in primary care centers Providers: pediatricians and nurses trained to perform motivational interview The interviews are structured as follows: First, checking the accomplishment of objectives to motivate the participant. Second, a specific topic per visit is explained to the participant. Third, a task related to the topic (i.e. to plan a weekly menu for the family) is given to be brought back at the next visit. 4th. Objectives about diet, weight & physical activity are defined to be accomplished until the next visit.
  Arms: Obemat2.0 Intervention Group
Other: Usual Clinical Practice — Lifestyle (diet and physical activity) Duration: 12 (+3) months Description: 1visit/month to the primary care centers. Providers: pediatricians & nurses. Children assigned to the control group receive the usual treatment conducted in primary care centers based on the Clinical Practice Guidelines on the Prevention and Treatment of Child and Adolescent Obesity [Spanish Ministry of Science and Innovation], 2009). At visits, the family receive recommendations to carry out a balanced diet, to provide a moderate energy reduction from the previous intake. An increase in physical activity, both in terms of leisure activity, as sports is advised.
  Other Names: Usual Reccomendations given at the pediatric consultations
  Arms: Control Group

SUMMARY:
Animal models and studies on small samples of obese adults have shown that gut microbial diversity and certain types of bacteria could predict the efficacy of the dietetic treatment to improve body mass index (BMI) and the components of metabolic syndrome (MetS). Gut microbiota could distinguish the obese with metabolic syndrome patient than that metabolically healthy. Dietetic therapy could induce changes in the microbiota that could lead to improvement of BMI and the components of the MetS. The aim of MICROBEkids is to test whether the motivational intervention a motivational intervention (OBEMAT2.0) (PI15/00970) is more effective than the conventional intervention to increase the gut microbial diversity and, as a consequence, to improve BMI and MetS components. The role of gut microbiota (through modulation of the short chain fatty acids) will be analyzed as cardiovascular risk factor and as predictor of treatment success. These objectives will be achieved through a clustered clinical trial design with an intervention group that will receive a motivational therapy compared to a control group that will receive a conventional intervention, both during 12 months. The study sample are 319 children (n= 167 in the intervention group) that were enrolled in the clinical trial OBEMAT2.0 (PI15/00970), have had a comprehensive clinical assessment before the intervention (ages 8 to 14) and after 12 months (+3) of therapy (ages 9 to 15) and furthermore have participated in a biological samples collection for the investigation on childhood obesity (COLOBEPED, reference C.0004585).

DETAILED DESCRIPTION:
The study will provide light to several hypothesis:

- The main hypothesis is that the dietetic intervention in obese children may improve the components of the metabolic syndrome by mediation (at least in part) of changes in the microbiota.

Other secondary hypothesis to be demonstrated are:

* The microbiota (before the treatment) could be a determinant factor of the metabolic syndrome (inflamation, serum lipid profile, insulin resistance) being a key feature differentiating the metabolically healthy obese from the obese with metabolic syndrome.
* A dietary pattern rich in vegetables and fruits is associated to a gut microbiota profile preventing the metabolic syndrome

How these hypothesis will be demonstrated? A motivational structured intervention to reduce weight is applied (under randomized clustered design) to obese children, that are compared to an active intervention (not structured) provided by health care professionals, both groups during 12 months (+3).

A baseline and final assessment (before and after the intervention) are performed, in which the following information is collected:

* Socioeconomics
* Anthropometry (weight, height, waist circumference) to calculate the obesity degree (BMI z- score) and the presence of abdominal obesity
* Body composition: deuterium dilution (in a subsample), bioimpedance, Dual X-Ray Absorptiometry and Air displacement pletismography (BodPod)
* Blood sample drawn: to analyze lipids profile and insulin resistance
* Fecal sample: the gut microbiota diversity and the presence of specific bacteria will be analyzed
* Dietary intake by a food frequency questionnaire: diet will be analyzed as dietary patterns
* Systolic and diastolic blood pressure (which will be adjusted as z-score)

ELIGIBILITY:
Inclusion Criteria:

* Age range between 8 and <14 years at enrolment (so that, children would end the treatment at maximum age of 15 years
* BMI > 97th percentile of Hernandez references from 1988 (Hernández et al., 1988) as indicated by the Guidelines for Clinical Practice of the Spanish Health System (Grupo de trabajo de la Guía de Práctica Clínica sobre la Prevención y el Tratamiento de la Obesidad Infantojuvenil. Ministerio de Ciencia e Innovación [Spanish Ministry of Sciencee and Innovation], 2009) for the diagnose of the childhood obesity.

Exclusion Criteria:

* Children with eating disorders
* Families not available to attend to scheduled visits
* Simultaneous participation in another clinical trial
* Presence of endocrine disorders (GH disorder, hypothyroidism, Cushing's disease, early puberty or other)
* Lack of command of local languages

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Fecal microbial diversity (diversity index like Gini-Simpson) | 12 (+3) months
  Effect of the intervention on increments of Fecal microbial diversity

SECONDARY OUTCOMES:
Fecal Short Chain Fatty Acids: butyrate acid (μg) | 12 (+3) months
  Effect of the intervention and microbiota on increments Short Chain Fatty Acids
Fecal Short Chain Fatty Acids: acetic acid (μg) | 12 (+3) months
  Effect of the intervention and microbiota on increments Short Chain Fatty Acids
Fecal Short Chain Fatty Acids: propionic acid (μg) | 12 (+3) months
  Effect of the intervention and microbiota on increments Short Chain Fatty Acids
Akkermansia Muciniphila (cfu) | 12 (+3) months
  Effect of the intervention on increments of Akkermansia Muciniphila in feces

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Luque, Principal Investigator — Institut d'Investigació Sanitària Pere Virgili
Locations (3):
- Spain (3):
  - Faculty of Medicine, C/ Sant Llorenç 21, Reus, Tarragona
  - Iispv- Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital de Tarragona Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alcazar M, Escribano J, Ferre N, Closa-Monasterolo R, Selma-Royo M, Feliu A, Castillejo G, Luque V; Obemat2.0 Study Group. Gut microbiota is associated with metabolic health in children with obesity. Clin Nutr. 2022 Aug;41(8):1680-1688. doi: 10.1016/j.clnu.2022.06.007. Epub 2022 Jun 15. PMID 35777107
- See also: Preliminar (baseline) results — https://pubmed.ncbi.nlm.nih.gov/35777107/